

Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

#### INFORMATION AND INFORMED CONSENT SHEET

| Title | MP3-pulses COVID-19. METHYLPREDNISOLONE PULSES VERSUS DEXAMETHASONE RECOVERY REGIMEN IN PATIENTS WITH PNEUMONIA DUE TO SARS-COV-2 CORONAVIRUS INFECTION |
|---|---|
| Protocol Code | MP3-pulses-COVID-19 |
| Principal Investigator | |
| Service | |

#### Introduction

We are writing to inform you about a research study in which you are invited to participate. Participation is voluntary. Please take the time to read the information below and refer to what you want. Ask the researcher in this study if anything is unclear to you or if you want to learn more.

As you know, he is hospitalized for a confirmed condition or very compatible with coronavirus infection.

This is still a poorly understood disease. So far, there is no treatment specifically directed against this virus. However, there are several medications that have been found to be effective in some patients. These treatments, and other general measures, are being administered to you, in a way that is tailored to your clinical situation.

After infection with the virus, the body's defense systems organize a response to try to eliminate it. That response sometimes leads to inflammation of some organs, especially the lungs. For this reason, medications, such as corticosteroids, are sometimes used in this disease to try to decrease the harmful part of the inflammation.

At the end of June 2020, a large clinical trial (RECOVERY) conducted by the British public health system was the first to clearly demonstrate that corticosteroids are useful in the management of this disease when patients notice shortness of breath and require supplemental oxygen. Since then, this treatment has been common in all patients with COVID-19 pneumonia.

However, even though we know the usefulness of corticosteroid treatment, we still need to know what the ideal dose and duration of treatment is and whether the use of higher doses could be even more beneficial for the patient.

#### Objective of the study

The aim of the study is to compare the effect of high-dose methylprednisolone boluses versus the dexamethasone intermediate-dose regimen (the one used in the RECOVERY trial) in COVID-19 patients with non-critical respiratory failure.



Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

This research study has been approved by the Ethics Committee for Research with Medicines of the Salamanca Health Area and is carried out in accordance with current legislation, Royal Decree 1090/2015 of 4 December and European Regulation 536/2014 of 16 April, which regulate clinical trials with medicines. and in accordance with the standards of good clinical practice.

#### **Study Procedures and Potential Risks and Discomforts**

The study will compare the outcome of a limited number of patients divided into 2 groups. Both groups will be treated with glucocorticoids. One of them at the dose tested in the RECOVERY trial for 10 days. The other group will receive higher doses, but for only three days, known as methylprednisolone boluses.

The study has been reviewed and approved by the appropriate committees in order to ensure its quality and the safety of the patients included.

During the study, your doctor will inform you of the need to receive steroid treatment. You will then be assigned to one of two study groups:

- 1) Group 1: dexamethasone 6 mg for 10 days, the first three intravenously and the rest either orally or intravenously depending on the patient
- 2) Group 2: 3 boluses of intravenous methylprednisolone. You will also continue with all other treatments indicated for your particular case.

This assignment will be made 1:1 randomly, you have an equal chance of getting one or the other treatment arm. In addition, the assignment is done centrally, so neither you nor the doctor know a priori the branch of treatment that you may have.

Your doctor will monitor your progress and may always modify the treatment, or cancel the study, if he or she considers it preferable in terms of your evolution. Subsequently, you will collect the main data from your story to analyze the results. That data will be encrypted, with no possibility of you being identified.

The rest of the treatment will be included in your hospital's COVID-19 management protocol. No diagnostic laboratory or imaging tests other than those that would normally be performed during the admission of a patient with COVID-19 infection will be performed. During admission, you will have at least 2 x-rays and 3 analysis determinations.

In addition, 28 days after the start of treatment, a follow-up visit will be made to see your progress, in which some more tests will be carried out, such as blood tests and imaging tests. Similarly, at 12 weeks or if you are removed from the study, of your own volition or by decision of your doctor, prematurely at any time during your participation, you will have another follow-up visit. This visit can be carried out in person or by phone, if the doctor and you consider it appropriate, so, in addition to asking you about your condition, you could be given some more tests such as blood tests and imaging tests if the visit is face-to-face.



Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

Given the current situation of the global health crisis, in the event of a lack of stock of any of the active ingredients in the study, it could be decided to use other glucocorticoid preparations in doses equivalent to that of methyl-prednisolone, according to the following table:

| Active ingredient | Guideline | Equivalence in<br>methyl-<br>prednisolona | Equivalence in prednisone |
|---|---|---|---|
| Dexamethasone | 6 mg/24h | 30 mg/24h | 37.5mg/24h |
| Methylprednisolona | 250mg/24h | N/A | 312.5 mg/24h |
| Hydrocortisone | 50-100mg/6h | 20-40 mg/12h | 25-50 mg/12h |

In both arms of the study, or in the case of administering any of the other glucocorticoid preparations, the risks inherent to the use of corticosteroids may appear, such as mainly the increased risk of infection added to the infection by the virus itself (rare), increased blood glucose levels (rare) or mood disorders (very rare). Other side effects of corticosteroids such as high blood pressure, dyslipidemia, diabetes or osteoporosis are not expected in this study given the short duration of treatment. Participation in this study would not cause any discomfort, and does not involve additional health risk.

If you do not agree to participate, your doctor will continue your current treatment and may eventually consider administering the 10-day dose of dexamethasone as well.

#### **Voluntary Participation and Withdrawal**

You are free to decide whether or not you want to take part in this study, participation is completely voluntary. If you choose to participate, you still have the ability to withdraw at any time, without explanation, and without any penalty or negative consequences for you. If you change your mind about your data, you have the right to request its destruction or anonymization, through your doctor/researcher. However, you should be aware that the data obtained in the analyses carried out up to that point may be used for the purposes requested and may be kept in compliance with the corresponding legal obligations.

If you do not participate in the study, you will receive treatment according to standard clinical practice, and there is even the possibility that, if your doctor decides to do so, you may receive one of the drugs offered in this study. If you want, the study doctor will give you more information.

#### **Potential Benefits**

You may not get any health benefits from taking part in this study. However, the information gained from this trial may contribute to medical progress and could help other patients suffering from their disease in the future.

You will not receive any financial benefit from the transfer of the data provided, nor will you have rights to possible commercial benefits from the discoveries that may be made as a result of the research carried out.



Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

#### Data protection and confidentiality

All information about your results will be treated as strictly confidential. Both the Centre and the Promoter are responsible for the processing of your data and undertake to comply with the data protection regulations in force, currently Organic Law 3/2018, of 5 December, on the Protection of Personal Data and Guarantee of Digital Rights and Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on Data Protection (GDPR). The data collected for the study will be identified by a code, so that no information that could identify you is included, and only the research team will be able to relate this data to you. The research team will analyse your data based on the legitimate interest of achieving the purposes of the study. Subsequently, your personal information will only be retained by the health care center and the research team for other scientific research purposes if you have given your consent to do so and if permitted by applicable law and ethical requirements.

If the results of the study are susceptible to publication in scientific journals, at no time will personal data of the participants in this research be provided. We inform you that you have the right to access, rectify or cancel your data, and you can limit the processing of data that is incorrect, request a copy or transfer to a third party of the data you have provided for the study. To exercise their rights, or in the event that the participant wishes to provide further information on the processing of their personal data, the principal investigator of the study whose details are specified at the end of this document may be contacted by the Data Protection Officer of the Regional Health Management (dpd@saludcastillayleon.es) or our centre (dpd.husa@saludcastillayleon.es). You also have the right to contact the Data Protection Agency if you are not satisfied.



Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

#### Information on results

At your request, at the end of the study and in accordance with article 27 of Law 14/2007 on Biomedical Research, you may be provided with information on the results of this research work.

| I authorize those responsible for the project to use my data for the purposes and in the manner described in this document. |
|---|
| □ IF □ NO |
| I consent to the future use of the data that have been collected in this research study to conduct other research related to the medical specialty or research area of this study |
| □ IF □ NO |
| I consent to my medical records being accessed again in the future to collect data that is considered important for other research related to the medical specialty or research area of this study |
| □ IF □ NO |

## **Contact details of the research team:**

If you have any questions or need more information, please contact:

Name:

Telephone:



Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

# **INFORMED CONSENT**

| Title | MP3-pulses COVID-19. METHYLPREDNISOLONE PULSES VERSUS DEXAMETHASONE RECOVERY REGIMEN IN PATIENTS WITH PNEUMONIA DUE TO SARS-COV-2 CORONAVIRUS INFECTION |
|---|---|
| Protocol Code | MP3-pulses-COVID-19 |
| Principal Investigator | |
| Service | |
| । (First and Last Name) | |
| I have read the informa | tion sheet that has been given to me about the study. |
| I've been able to ask qu | estions about the study. |
| I have received enough | information about the study. |
| I have spoken with the | nvestigator |
| I understand that my pa | articipation is voluntary. |
| I understand that I can | withdraw from the study: |
| 1º Whenever yo | ou want |
| 2º Without hav | ing to give explanations |
| 3º Without hav | ing any negative repercussions |
| | participate in the clinical trial and authorize the use of all information that I will receive a signed copy of this informed consent. |
| Participant's signature | Date |



Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

# **INFORMED CONSENT IN THE PRESENCE OF A WITNESS\***

| Title | MP3-pulses COVID-19. METHYLPREDNISOLONE PULSES VERSUS DEXAMETHASONE RECOVERY REGIMEN IN PATIENTS WITH PNEUMONIA DUE TO SARS-COV-2 CORONAVIRUS INFECTION |
|---|---|
| Protocol Code | MP3-pulses-COVID-19 |
| Principal Investigator | |
| Service | |
| (Patient's name and sur | rname) |
| । (Name and Surname o | f Witness) |
| · | ent has read (or has been read to them if they are unable to do so on tion sheet that has been given to them about the study. |
| He was able to ask ques | tions about the study. |
| You have received enou | igh information about the study. |
| Have you spoken with t | he Investigator |
| You understand that yo | ur participation is voluntary. |
| You understand that yo | u may withdraw from the study: |
| 1º Whenever yo | ou want |
| 2º Without having to give explanations | |
| 3º Without havi | 3º Without having any negative repercussions |
| , - | o participate in the clinical trial and authorize the use of all information nd that you will receive a signed copy of this informed consent. |
| Signature of the witness Date | S |

Researcher's name and signature



Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

\*When the patient is unable to sign and gives oral consent. The witness may be a family member or healthcare worker.

## **INFORMED CONSENT FOR LEGAL REPRESENTATIVE**

| Title | | MP3-pulses COVID-19. METHYLPREDNISOLONE PULSES VERSUS DEXAMETHASONE RECOVERY REGIMEN IN PATIENTS WITH PNEUMONIA DUE TO SARS-COV-2 CORONAVIRUS INFECTION | | | | |
|---|---|---|---|---|---|---|
| Prot | ocol Code | МР3-рі | MP3-pulses-COVID-19 | | | |
| Princ | cipal Investigator | | | | | |
| Serv | ice | | | | | |
| (Patie | ent's name and su | ırname) | | | | |
| I | (Name | and | Surname | of | Legal | Representative) |
| I have | e read the inform | ation shee | t that has been gi | ven to me | about the stud | y. |
| He wa | as able to ask que | estions abo | out the study. | | | |
| You h | ave received eno | ugh inforn | nation about the s | study. | | |
| Have | you spoken with | the Invest | igator | | | |
| I unde | erstand that your | participat | ion is voluntary. | | | |
| I unde | erstand that you | may withd | raw from the stud | ły: | | |
| | 1º Whenever y | ou want | | | | |
| | 2º Without ha | ving to give | e explanations | | | |
| | 3º Without ha | ving any ne | egative repercussi | ons | | |
| | , - | | e in the clinical tr<br>vill receive a signe | | | e of all information<br>onsent. |
| Signa | ture of the legal r | epresenta | tive | | | Date |
| Resea | rcher's name and | d signature | <u> </u> | | | Date |



Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

# **INFORMED CONSENT IN THE PRESENCE OF A WITNESS\***

| Title | MP3-pulses COVID-19. METHYLPREDNISOLONE PULSES VERSUS DEXAMETHASONE RECOVERY REGIMEN IN PATIENTS WITH PNEUMONIA DUE TO SARS-COV-2 CORONAVIRUS INFECTION |
|---|---|
| Protocol Code | MP3-pulses-COVID-19 |
| Principal Investigator | |
| Service | |
| (Patient's name and sur | name) |
| । (Name and Surname o | f Witness) |
| · | ent has read (or has been read to them if they are unable to do so on tion sheet that has been given to them about the study. |
| He was able to ask ques | tions about the study. |
| You have received enou | gh information about the study. |
| Have you spoken with the | he Investigator |
| You understand that yo | ur participation is voluntary. |
| You understand that yo | u may withdraw from the study: |
| 1º Whenever yo | ou want |
| 2º Without having to give explanations | |
| 3º Without havi | 3º Without having any negative repercussions |
| · - | o participate in the clinical trial and authorize the use of all information and that you will receive a signed copy of this informed consent. |
| Signature of the witness | <u> </u> |

Date



Researcher's name and signature

EudraCT: 2020-005026-28

Sponsor: Instituto de Investigación Biomédica de Salamanca (IBSAL)

## **REVOCATION OF CONSENT**

| Title | MP3-pulses COVID-19. METHYLPREDNISOLONE PULSES VERSUS DEXAMETHASONE RECOVERY REGIMEN IN PATIENTS WITH PNEUMONIA DUE TO SARS-COV-2 CORONAVIRUS INFECTION | | | | |
|---|---|---|---|---|---|
| Protocol Code | MP3-pulses-COVID-19 | | | | |
| Principal Investigator | | | | | |
| Service | | | | | |
| D/Dña | | | | | |
| l voluntarily | revoke | the | consent | given | on |
| | | | | | _ |
| Participant's signature | | | | | Date |